CLINICAL TRIAL: NCT00246883
Title: Effect of Regular Exercise on Vascular Function and Cardiovascular Risk in a Sedentary Work Force: The NHLBI "Keep the Beat" Program
Brief Title: Effect of Regular Exercise on Vascular Function and Cardiovascular Risk in a Sedentary Work Force
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060018; 06-H-0018
Record Dates: First submitted 2005-10-29; First posted 2005-10-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-15

CONDITIONS: Vascular Formation
Keywords: Endothelial Progenitor Cells; Nitric Oxide; Brachial Artery Reactivity; Physical Fitness; C-reactive Protein; Exercise; Vascular Function
MeSH Terms: conditions — Motor Activity | interventions — Exercise

INTERVENTIONS:
Procedure: Exercise

SUMMARY:
This study will evaluate the effects of NHLBI's employee exercise program, Keep the Beat, on blood vessel function. Damage to blood vessels can cause narrowing of the vessels, resulting in reduced blood flow to parts of the body such as the heart. Stem cells called endothelial progenitor cells, or EPCs, may be able to heal blood vessel damage. Exercise, such as walking on a treadmill, can help move EPCs from the bone marrow where they originate into the blood stream to help heal the damaged blood vessels. The Keep the Beat program encourages NHLBI employees to exercise 15 minutes during the workday and provides exercise facilities to accomplish this.

NHLBI employees who have access to NIH exercise facilities may be eligible for this study. Candidates must have no history of heart disease, must not currently be exercising more than 1.5 hours per week and must not have participated in the Keep the Beat program for 3 months prior to entering the study. They are screened with blood tests and blood pressure measurements.

Participants undergo the following tests and procedures before beginning the study and 3 months after participating in Keep the Beat:

* Blood tests to identify EPCs and their function, measure the level of nitric oxide (a gas produced by healthy blood vessels), and measure C-reactive protein (an inflammatory marker that may be a risk factor for cardiovascular disease).
* Brachial artery reactivity study to measure how well the arteries widen. An ultrasound device is placed over the subject's artery just above the elbow. The device measures the size of the artery and the flow of blood through it before and after a pressure cuff is inflated around the forearm.
* Treadmill exercise testing to evaluate physical fitness. Subjects exercise on a treadmill for as long as they can. An exercise specialist is present throughout the test. Heart rhythm and oxygen saturation are monitored continuously and blood pressure is measured every 3 minutes.

DETAILED DESCRIPTION:
Evidence suggests that Americans are becoming increasingly sedentary at work and at home due to technological advances. Physical inactivity coupled with excess caloric intake, especially of calorie-rich fast foods, are responsible for the epidemic of obesity in this country. Physical inactivity in obese and non-obese individuals increases the risk of cardiovascular disease and all-cause mortality. Premature cardiovascular disease leads to lost productivity in the work place, impaired quality of life, and escalating health care costs. In response to these concerns, the American Heart Association advocates 30 minutes of aerobic exercise most days; however, busy schedules coupled with a lack of convenient access to exercise equipment (or motivation to use it) limit adoption of regular exercise by many. One year ago, the National Heart, Lung, and Blood Institute (NHLBI) initiated the Keep the Beat program which encourages Institute employees to engage in fifteen minutes of exercise during the work day, and provides exercise equipment at specific work sites to accomplish this goal. Yet, fewer than 10% of NHLBI employees regularly participate in Keep the Beat and many who initially enrolled have failed to continue participation. The purpose of our prospective cohort study is to determine whether participation in the Keep the Beat program can improve an important measure of cardiovascular risk-arterial endothelial function-by stimulating bone marrow-derived endothelial progenitor cells to repair endothelium. We propose to characterize important components of vascular health by measuring endothelial nitric oxide bioactivity, as determined by brachial artery reactivity to shear stress and nitric oxide metabolites in blood, and vascular repair potential, as determined by endothelial progenitor cell number and function, at baseline and at 3 months in National Institutes of Health employees who agree to participate in Keep the Beat. Secondary analyses will include other biomarkers of risk, such as C-reactive protein, blood pressure, body mass index, lipid profile, fasting glucose/insulin, and homeostasis model assessment index, to be measured in our study and subgroup analyses of participants at particularly high cardiovascular risk (greater than 20% over 10 years), minorities, and women. Demonstration of improved vascular function, with implications of reduced cardiovascular risk, may serve as an incentive for greater employee participation in established employer-initiated programs, and for adoption of similar programs by other employers. If objective benefit cannot be demonstrated in vascular function and other biomarkers of risk, modification of the program may be required to reduce cardiovascular risk.

ELIGIBILITY:
* INCLUSION CRITERIA:

Employees of NHLBI who are not currently participating in the Keep the Beat program (this may include employees who have previously registered for Keep the Beat program, but who have not participated in the past 3 months) and NIH employees who can use the excercise rooms in Building 10, Building 31, or Rockledge II.

No medical condition that might prohibit safe participation in the Keep the Beat program.

Subject understands protocol and provides written, informed consent in addition to willingness to comply with specified follow-up evaluations.

EXCLUSION CRITERIA:

Heart disease as indicated by history of myocardial infarction, documented disease on coronary angiography, coronary artery stent placement, congestive heart failure, significant structural heart disease (e.g. hypertrophic or dilated cardiomyopathy, or valvular heart disease), or positive treadmill exercise test at baseline.

Baseline blood pressure systolic greater than 140 mmHg or diastolic greater than 90 mmHg on 2 measures with or without hypertensive medications. Subjects will be encouraged to seek evaluation by their primary care provider.

Baseline fasting blood glucose greater than 126 mg/dl, if subject previously undiagnosed as being diabetic. Subjects will be encouraged to seek evaluation by their primary care provider.

Baseline fasting LDL greater than 190 mg/dl. Subjects will be encouraged to seek evaluation by their primary care provider.

Physically unable to perform the Keep the Beat program due to neurologic or orthopedic conditions.

Pregnant women will be excluded due to large hormonal changes in pregnancy that affect study variables and potential pregnancy-related restrictions on exercise.

Subjects currently exercising more than 1.5 hours per week including brisk walking, sporting activities (such as basketball), and other deliberate exercise.

Subjects may not be currently participating or participate over the course of the study in another study protocol which includes blood draws or interventions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2005-10-26; Study Completion 2009-04-15

PRIMARY OUTCOMES:
Improvement in brachial artery dilator responsiveness to shear stress as a bioassay for endothelium-dependent nitric oxide bioavailability following 3 months participation in the Keep the Beat program as compared with baseline measuraements.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Blair SN, Kohl HW, Gordon NF, Paffenbarger RS Jr. How much physical activity is good for health? Annu Rev Public Health. 1992;13:99-126. doi: 10.1146/annurev.pu.13.050192.000531. PMID 1599603
- [Background] Hu G, Tuomilehto J, Silventoinen K, Barengo NC, Peltonen M, Jousilahti P. The effects of physical activity and body mass index on cardiovascular, cancer and all-cause mortality among 47 212 middle-aged Finnish men and women. Int J Obes (Lond). 2005 Aug;29(8):894-902. doi: 10.1038/sj.ijo.0802870. PMID 15724141
- [Background] Brownson RC, Boehmer TK, Luke DA. Declining rates of physical activity in the United States: what are the contributors? Annu Rev Public Health. 2005;26:421-43. doi: 10.1146/annurev.publhealth.26.021304.144437. PMID 15760296